CLINICAL TRIAL: NCT05313464
Title: Effect of Parental Enteral Nutrition on Quality Of Parent-Child Interactions: Prospective Randomized Monocentric Study (PREMIAM)
Brief Title: Effect of Parental Enteral Nutrition on Quality Of Parent-Child Interactions
Acronym: PREMIAM
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Collaborators: Le Laboratoire de Psychopathologie et Processus de Santé (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PREMIAM
Record Dates: First submitted 2022-02-04; First posted 2022-04-06 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Premature; Parent-Child Relations
Keywords: Premature; child at 32 of gestational age; enteral nutrition; skin to skin; push on syringe pump; Parent-Child Relations
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nutrition pushed by parents (Experimental): enteral nutrition pushed by parents
  Interventions: Other: parent-pushed enteral feeding
- syringe pump (Active Comparator): Enteral nutrition with syringe pump
  Interventions: Other: syringe-push enteral feeding

INTERVENTIONS:
Other: parent-pushed enteral feeding — skin-to-skin enteral nutrition pushed by the parent
  Arms: nutrition pushed by parents
Other: syringe-push enteral feeding — skin to skin nutrition with syringe pump
  Arms: syringe pump

SUMMARY:
Studies underline both the importance of the link and contact that occurs in the earliest days of life and the need to involve parents early with their premature child.

However, the impact of parental nutrition on the later active nutrition and on the quality of parent-child interactions is currently unknown.

PREMIAM study investigates whether active parental participation in enteral nutrition improves the interactions between the infant and his parents, making them more sensitive to their baby's signals and promoting their relational adjustment.

DETAILED DESCRIPTION:
The importance of parental participation in the feeding of preterm infants has been highlighted by Gianni. In his study of 81 preterm infants in the tertiary centre , the early parental bottle feeding and the skin-to-skin contact were factors promoting withdrawal from enteral nutrition. Moreover, actively participate in care even complex, is desired by parents.

Recently, a study compared 10 parent-child dyads and showed that enteral nutrition pushed by a parent (parental nutrition, NP) in comparison of the electric syringe pump , allowed a better perception of the tube by the parents and gave them a sense of utility. The same team randomized 17 preterm infants, born after 28 WA( week amenorrhoea), to receive or not à parent-pushed enteral nutrition The child's behavior changes during nutrition were analyzed in both arms, after scoring of the videos feeding according to the NICAP® ( individualized neonatal assessment and developmental care program) method. Signs of well-being and relaxation of members were more present in case of parental involvement in the delivery of nutrition. These preliminary studies suggest that parental nutrition is well tolerated and improves the comfort of the child and parent during nutrition.

However, the impact of parental nutrition on the subsequent active nutrition and on the quality of parent-child interactions is currently unknown.

ELIGIBILITY:
Inclusion Criteria:

Children born before 30 SA Age of child at start of study: 32 SA

Exclusion Criteria:

* Child with ongoing infection, neurological pathology More than one desaturation and/or bradycardia per hour within 12 last hours Balloon ventilation in last 12 hours
* Medical contraindication to oral nutrition
* Intubated child
* Parents with a disabling mental illness
* Parents not available
* Minor parents
* Parents under guardianship or protection of justice
* Refusal to sign consent
* Parents not affiliated with a social security system

Ages: 30 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2022-04-15 (Actual); Primary Completion 2027-04-15 (Estimated); Study Completion 2027-12-28 (Estimated)

PRIMARY OUTCOMES:
behavioural interactions (visual, vocal, mimic) | 34 (W) weeks of gestational age
  interactions during the first 10 minutes of an interactive sequence of a premature in the arms of his parent, filmed and coded with The Observer XT software to 34 WA, starting from 3 behaviors of the premature: vocalization, face look mother" and smile

SECONDARY OUTCOMES:
Mother and Father Self-Question Assessment of Parental Competence: The Cognitive and Parental Behaviour Scale (PACOTIS) | at Month 4
  Parents indicate on an eleven point scale (0 = not at all what I think, feel, or do; 10 = exactly what I think, feel, or do) to what extent each statement accurately describes their actions, thoughts or feelings in the context of interacting with their infants. The parental self-efficacy (6 items, α = .82), and perceived parental impact (5 items, α = .68) subscales include statements relating to beliefs about parenting competence and their impact on the child, while the parental hostile-reactive behaviours (7 items, α = .73), parental overprotection (5 items, α = .60), and parental warmth (5 items, α= .78) subscales assess parents' involvement in different types of behaviour with their child.
  Scores from each subscale are averaged out of 10; higher scores indicating greater use of these behaviours. the Perceived parental impact subscale items are reverse coded.
Edinburgh Postpartum Depression Risk Rating Scale (EPDS) | at inclusion, at 32, 34 and 37 weeks of gestation
  Questionnaire EPSD QUESTIONS 1, 2, & 4 (without an *) Are scored 0, 1, 2 or 3 with top box scored as 0 and the bottom box scored as 3.
  QUESTIONS 3, 5-10 (marked with an *) Are reverse scored, with the top box scored as a 3 and the bottom box scored as 0.
  Maximum score: 30 Possible Depression: 10 or greater Always look at item 10 (suicidal thoughts)
Parental Stressor Scale: Neonatal Intensive Care Unit (PSS: NICU) | at 32, 34, and 37 weeks of gestation
  The scale consists of four subscales that measure stress related to (a) the sights and sounds of the unit (5 items), (b) the appearance and behaviours of the infant (19 items), (c) the impact on the parents' role and their relationship with their baby (10 items), and (d) the staff behaviours and communications (11 items). There is also a general stress-level question that summarizes the parents' overall feeling of stress related to having an infant in the NICU.
  The responses to the PSS: NICU were scored on a 5- point Likert scale from 0 to 5 where 0 means no experience at all with the situation or phenomenon, 1 (not at all stressful) to 5 (extremely stressful).
  Mean scores and standard deviation were obtained for each subscale and total scale separately for mothers and fathers and the overall stress scores was then calculated. Parental stress levels were classified according to the points on Likert scale as low (1-1.9), moderate (2-3.9) and high (4-5).
Number of desaturation | every day betwenn 32 and 34 weeks of gestation
  Number of desaturation
Number of vomiting | every day between 32 and 34 weeks of gestation
  Number of vomiting
Exit age on return home | through study completion, an average of 41 week of gestation
  age of the infant when leaving the hospital
Parental time in hours | at 34 week of gestation and 37 week of gestation, calculated over 7 days
  time spend withe child
Number of meals and baths given by parents | from 32 week of gestation to 37 week of gestation
  Number of meals and baths given by parents
Duration of transition from passive to active feeding in number of days | from 32 week of gestation to 37 week of gestation
  Duration of transition from passive to active feeding in number of days
Average duration (minutes) of feeding/feeding | at 37 week of gestation
  Average duration (minutes) of feeding/feeding
Number and duration of skin-to-skin sessions in minutes | from inclusion to exit of service ( up to 45 week of gestation)
  Number and duration of skin-to-skin sessions in minutes
Duration of breastfeeding in number of days. | from 32 week of gestation to 37 week of gestation
  Duration of breastfeeding in number of days.
Number of children with infant formula change | between 32 week of gestation and 37 week of gestation
  Number of children with infant formula change
Evolution of the Z-weight score | 32 week of gestation at the exit of the child.
  The score shows the standard deviation above or below the mean on the growth chart. If you have looked at a growth chart of a patient or your own child, you will recall it contains curve shaped lines with various percentiles on it.
  The middle line is the 50th%Ile and they extend out to the 97%ile percentile and 3rd%Ile. So, a z score of 0 is the equivalent of the 50th%ile or average of what you are measuring (weight, height, weight for height or BMI) for that age.
  A z score of +1 means your plots fall at the 15th%ile or 85th%Ile and a z score of +2 falls roughly at the 3rd or 97%Ile. z scores run positively (+1. +2.+3) or negatively (-1, -2. -3) and so on.
Brunet-Lézine and Neurological Evaluation of Amiel Tison simplified by a psychomotor specialized in the development of premature babies to assess the psychomotor development of infants at | 4 months of age corrected.
  It may apply from the first month up to 5 years. It includes observations on posture, coordination, language, social-personal conduct.
  The Brunet-Lézine scale was developed by Odette Brunet and Irene Lézine. It provides a development quotient (Q.D.).
The Montreal Children's Hospital Feeding Scale [MCH-Feeding Scale] | 4 months of age corrected
  scale for identification of feeding problems. The final scale consisted of 14 items covering the following feeding domains with some overlap: oral motor (items 8 and 11), oral sensory (items 7 and 8) and appetite (items 3 and 4). Other items covered maternal concerns about feeding (items 1, 2 and 12), mealtime behaviours (items 6 and 8), maternal strategies used (items 5, 9 and 10) and family reactions to their child's feeding (items 13 and 14).
  Each item is rated on a seven-point Likert scale with anchor points at either end. Seven items are scored from the negative to positive direction, and the other seven from the positive to negative direction. The primary feeder marks each item according to frequency or difficulty level of a particular behaviour or the level of parental concern. The total feeding problem score is obtained by adding the scores for each item after reversing the scores of seven items from negative to positive
Number bradycardia | every day betwenn 32 and 34 weeks of gestation
  Number bradycardia

CONTACTS AND LOCATIONS:
Overall Officials: Nelly THOMAS, Principal Investigator — Centre Hospitalier Intercommunal Créteil
Locations (1):
- Centre Hospitalier Intercommunal Créteil, Créteil, Val-deMarne, France

IPD SHARING:
Plan to Share IPD: No